CLINICAL TRIAL: NCT01770080
Title: Efficacy and Safety of Euminz® (10% Ethanolic Solution of Peppermint Oil for Topical Use) Compared to Placebo in Patients With Episodic Tension-type Headache (ETTH); Phase IV Clinical Trial
Brief Title: Efficacy of Euminz® for Tension-Type Headache
Acronym: CAS/B/016611
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Cassella-med GmbH & Co. KG (Industry)
Responsible Party: Principal Investigator, Rainer Stange, Dr. med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011-004777-89
Record Dates: First submitted 2013-01-09; First posted 2013-01-17 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Episodic Tension-Type Headache
MeSH Terms: interventions — peppermint oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Euminz® (Active Comparator): Acute treatment (3 to 5 time topical use of Euminz® = 10%ethanolic solution of peppermint oil) will start immediately after assessment of a baseline pain intensity of at least moderate pain (3 on VPRS).
  Interventions: Drug: Euminz®
- Placebo (Placebo Comparator): Acute treatment (3 to 5 time topical use of Placebo= 0,5% ethanolic solution of peppermint oil) will start immediately after assessment of a baseline pain intensity of at least moderate pain (3 on VPRS).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Euminz® — 3 to 5 time topical use of study drug.
  Other Names: Peppermint oil (10% ethanolic solution).
  Arms: Euminz®
Drug: Placebo — 3 to 5 time topical use of study drug.
  Other Names: Peppermint oil (0,5% ethanolic solution).
  Arms: Placebo

SUMMARY:
Efficacy and safety of Euminz® (10% ethanolic solution of peppermint oil for topical use) compared to placebo in patients with episodic tension-type headache (ETTH).

Prospective, double-blind, placebo-controlled, phase IV clinical trial; Parallel-groups design; Randomisation 1:1; First attack per patient will be evaluated for primary objectives, following attacks during study duration will be observed and documented.

Study duration per patient: 10 weeks

DETAILED DESCRIPTION:
To demonstrate the efficacy of Euminz® to reduce the intensity of headache symptoms experienced by patients with episodic tension-type headache. The two primary objectives will be tested hierarchically (a-priory ordered) to avoid alpha-adjustment:

First primary objective of the first headache episode is "pain-free" (0 or 1) after 2 hours measured on a six-step verbal pain rating scale (VPRS). Acute treatment (3 to 5 time topical use of Euminz®) will start immediately after assessment of a baseline pain intensity of at least moderate pain (3 on VPRS).

Second primary objective of the first headache episode will be the decrease of intensity of pain measured by a visual analogue scale (VAS). The difference from measure point 0 (before first application of Euminz®) on the VAS in comparison to 15, 30, 45, 60, 90 and 120 minutes after start of treatment will be shown as area under the curve representing the pain intensity difference (PID).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients from 18 years onwards
* History of ETTH for at least one year. The number of days with such a headache is ≥2 per month
* Onset of TTH below 65 years of age
* At least 10 previous headache attacks fulfilling the following four inclusion criteria:
* Patients with headache attacks lasting from 30 minutes to 7 days
* At least two of the following pain characteristics are present:
* - Pressing or tightening (non-pulsating) quality
* - Intensity of pain: moderate = unable to ignore (pain may inhibit, but does not prohibit activities)
* - Bilateral location
* - No aggravation by walking stairs or similar routine physical activity
* Headache is not accompanied by nausea or vomiting (anorexia may occur)
* Headache is not accompanied by a combination of the following symptoms: photophobia and phonophobia (only one may be present)
* 3 months retrospective history
* Willingness and ability to keep the patient's diary and to comply with the procedures of the study
* Written informed consent

Exclusion Criteria:

* Headaches other than TTH: (e.g. migraine, cluster headache, hypertension headache, drug-related headache,analgesic-induced headache,post-traumatic headache; associated migraine attacks are permitted if they are well recognized by the patient and if their frequency during the preceding year has not exceeded one per month)
* Presence of oromandibular dysfunction
* History of facial or cranial surgery
* Use of prophylactic drugs for headache within one month prior to enrolment
* Use of drugs for acute TTH treatment for ≥ 10 days of headache per month
* Anticipated problems in adhering to the self-observation procedure (e.g. because of work)
* Abuse of alcohol, narcotics or other drugs
* Serious illnesses within the last 3 months (e.g. myocardial infarction, cardiac insufficiency NYHA III and IV, low blood pressure, cerebral insult, diabetes mellitus, neuropathy, changes in the skin or neoplasms in the head)
* Epilepsy
* Intake of anti-psychotic, anti-depressant or anti-epileptic medication during the previous month
* Intake of long-acting non-steroidal anti-inflammatory drugs within the last month
* Planned start of new pharmacological or non-pharmacological therapies
* Any significant skin condition affecting face or neck
* Known hypersensitivity towards peppermint oil
* Previous use of Euminz® or any other essential oil solutions for headache in the last three months
* Participation in another clinical trial within the last month
* Accommodation in an institution at judicial or official request

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2013-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
First primary objective of the first headache episode is "pain-free" (0 or 1) after 2 hours measured on a six-step verbal pain rating scale (VPRS). | 2 hours
  Acute treatment (3 to 5 time topical use of Euminz®) will start immediately after assessment of a baseline pain intensity of at least moderate pain (3 on VPRS).

SECONDARY OUTCOMES:
Further headache attacks will be documented and evaluated during study duration (VPRS, VAS) and described as sum of pain intensity differences (SPID) | 10 weeks

OTHER OUTCOMES:
Safety | 48 hours
  Physical eximanations, overall assessments both by the patients and the investigator, vital signs, adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Yatin Shah, MD, Study Director — Charite University, Berlin, Germany
Locations (1):
- Charité, Chair of Complementary and Integrative Medicine, Berlin, State of Berlin, Germany